CLINICAL TRIAL: NCT03728608
Title: Optimal Feeding Tube Dwell Time in VLBW Infants to Reduce Feeding Tube Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB201700398 -N-A; R01NR016964-01A1 (NIH); 5KL2TR001429 (NIH); 5R01NR016964-04 (NIH)
Record Dates: First submitted 2018-10-24; First posted 2018-11-02 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Infection
Keywords: neonatal intensive care unit (NICU); feeding tube contamination
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1--Short Dwell (Active Comparator): Premature VLBW (very low birth weight) male and female infants will be randomly assigned to have their feeding tubes removed at 0-48 hours for the first 4 weeks of life.The feeding tube lumen, interluminal liquid and hub will be analyzed for level of contamination.
  Interventions: Device: Feeding tube dwell time of 48 hours
- Group 2--Long Dwell (Active Comparator): Premature VLBW (very low birth weight) male and female infants will be randomly assigned to have their feeding tubes removed at 7 days for the first 4 weeks of life.The feeding tube lumen, interluminal liquid and hub will be analyzed for level of contamination.
  Interventions: Device: Feeding tube dwell time of 7 day

INTERVENTIONS:
Device: Feeding tube dwell time of 48 hours — Feeding tube dwell time of 48 hours for first 4 weeks of life.
  Arms: Group 1--Short Dwell
Device: Feeding tube dwell time of 7 day — Feeding tube dwell time of 7 days for first 4 weeks of life.
  Arms: Group 2--Long Dwell

SUMMARY:
The study team will determine whether a decreased feeding tube dwell time will reduce feeding tube contamination

DETAILED DESCRIPTION:
Contaminated feeding tubes can occur in the neonatal intensive care unit (NICU) and have been associated with significant morbidity. Due to an immature immunologic systems, premature infants are at significant risk of complications related to contaminated feeding tubes. Feeding tube dwell time may affect the level of contamination. This study will determine if a maximum feeding tube dwell time of 48 hours reduces contamination compared to a maximum feeding tube dwell time of 7 days, thereby improving neonatal health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* be born to a mother who is at least 18 years of age and English or Spanish speaking
* born at < or equal to 30 weeks
* have a birthweight < or equal to 1500 grams
* be born to a mother who is COVID Negative
* have a feeding tube placed within 24 hours of birth
* be expected to require a feeding tube for 4 weeks following birth.

Exclusion Criteria:

* infant with known congenital GI anomalies
* infants which are not expected to live
* infants will be withdrawn from the study if they require abdominal surgery for GI morbidities

Ages: 30 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Parker, Principal Investigator — University of Florida
Locations (1):
- Unversity of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Started | 76 | 75
Completed | 58 | 62
Not Completed | 18 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 76 | 75 | 151
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks gestation] | 27.8 (2.19) | 27.3 (2.2) | 27.5 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 84
  Male | 32 | 35 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 34 | 60
  White | 41 | 37 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 76 | 75 | 151

OUTCOME MEASURES:

1. Primary Outcome: Amount of Contamination
Description: prepared solution of sectioned feeding tubes will be plated on Agar. After 24 hrs of incubation, unique colony types will be counted.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Colony forming units
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 58 | 62
Colony forming units | 357,000,000 (136,000,000) | 4,820,000,000 (1,860,000,000)

2. Secondary Outcome: Gastrointestinal Inflammation - S100A12
Description: The samples will be analyzed for inflammatory markers using S100A12. Values will be log10 transformed
Time Frame: 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 mg/dL
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
log10 mg/dL | 0.87 [0.72 to 1.01] | 0.98 [0.94 to 1.12]

3. Secondary Outcome: Gastrointestinal Inflammation - Calprotectin
Description: The samples will be analyzed for inflammatory markers using calprotectin immunoassays. Levels will be log10 transformed
Time Frame: 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 mg/dL
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
log10 mg/dL | 2.6 [2.5 to 2.7] | 2.6 [2.5 to 2.7]

4. Secondary Outcome: Hours of Parenteral Nutrition
Time Frame: 4 weeks
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
hours | 195.5 [165.5 to 230.8] | 196.4 [163.1 to 236.6]
Statistical Analysis 1: Comparison: Group 1--Short Dwell vs Group 2--Long Dwell; Test type: Superiority; p = 0.92, survival analysis

5. Secondary Outcome: Days With a Central Venous Line
Time Frame: 4 weeks
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
days | 236.7 [191 to 293.2] | 248.3 [193.3 to 318.8]
Statistical Analysis 1: Comparison: Group 1--Short Dwell vs Group 2--Long Dwell; Test type: Superiority; p = 0.65, survival analysis

6. Secondary Outcome: Length of Neonatal Intensive Care Stay
Time Frame: birth until discharge from the neonatal intensive care unit
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
days | 75.6 [70 to 81.7] | 75.8 [69.1 to 83.1]
Statistical Analysis 1: Comparison: Group 1--Short Dwell vs Group 2--Long Dwell; Test type: Superiority; p = 0.96, survival analysis

7. Secondary Outcome: Days to Reach Full Feeds
Time Frame: 4 weeks
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
days | 9.3 [8.5 to 10.1] | 9.4 [8.4 to 10.5]
Statistical Analysis 1: Comparison: Group 1--Short Dwell vs Group 2--Long Dwell; Test type: Superiority; p = 0.77, survival analysis

8. Secondary Outcome: Number of Infants With Necrotizing Enterocolitis
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
Participants | 4 | 6
Statistical Analysis 1: Comparison: Group 1--Short Dwell vs Group 2--Long Dwell; Test type: Superiority; p = 0.43, Regression, Logistic

9. Secondary Outcome: Number of Infants With Late Onset Sepsis
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
Participants | 19 | 21
Statistical Analysis 1: Comparison: Group 1--Short Dwell vs Group 2--Long Dwell; Test type: Superiority; p = 0.97, Regression, Logistic

10. Secondary Outcome: Episodes of Abdominal Distension
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
Participants | 21 | 22
Statistical Analysis 1: Comparison: Group 1--Short Dwell vs Group 2--Long Dwell; Test type: Superiority; p = 0.97, Regression, Logistic

11. Secondary Outcome: Number of Infants With a Direct Bilirubin > 2 mg/dL
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
Number analyzed (Participants) | 76 | 75
Participants | 5 | 5
Statistical Analysis 1: Comparison: Group 1--Short Dwell vs Group 2--Long Dwell; Test type: Superiority; p = 0.79, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Group 1--Short Dwell | Group 2--Long Dwell
All-Cause Mortality (participants affected / at risk) | 7/76 | 6/75
Serious Adverse Events (participants affected / at risk) | 21/76 | 22/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1--Short Dwell (N=76) | Group 2--Long Dwell (N=75)
Abdominal surgery (Gastrointestinal disorders) | 2 | 2
necrotizing enterocolitits (Gastrointestinal disorders) | 4 | 6
Late onset sepsis (Infections and infestations) | 19 | 21
abdominal distension (Gastrointestinal disorders) | 21 | 22
direct bilirubin greater than 2 mg/dl (Gastrointestinal disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT03728608/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03728608/ICF_001.pdf